CLINICAL TRIAL: NCT05986487
Title: Impact of Sleep-Disordered Breathing Management in Systemic Hypertension Control: METASLEEP Project
Status: Recruiting | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Ferran Barbe, Chair Respiratory Medicine, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: PMP22/00030
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Obstructive Sleep Apnea
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2 tubes EDTA (6 ml)
  * 2 tubes with separating gel for serum (6 ml)
  * 1 tempus RNA tube (2,5 ml)
  * 1 tube for urine and urine sediment (3 ml)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with nocturnal hypertension and/or non-dipper pattern and diagnosed with OSA: Patients with nocturnal hypertension and/or non-dipper pattern who undergo a sleep test, obtaining the diagnosis of obstructive sleep apnea, will be treated following the clinical practice standards.
  Interventions: Device: CPAP or usual practice; Device: Monitoring and intervention in follow-up
- Patients with nocturnal hypertension and/or non-dipper pattern and without OSA: Patients with nocturnal hypertension and/or non-dipper pattern undergoing a sleep test, the result of which is negative for obstructive sleep apnea disease.
  Interventions: Device: Monitoring and intervention in follow-up

INTERVENTIONS:
Device: CPAP or usual practice — CPAP (continuous positive airway pressure) is a machine that uses mild air pressure to keep breathing airways open while you sleep.
  Groups: Patients with nocturnal hypertension and/or non-dipper pattern and diagnosed with OSA
Device: Monitoring and intervention in follow-up — Each participating center can incorporate monitoring and intervention in the follow-up of patients into their work dynamics. Through the use of mobile applications, you can monitor the variables of: weight, diet, lifestyle, exercise and sleep. This intervention will help the patient to improve in different aspects of their health.

SUMMARY:
Hypertension is a frequent condition affecting 11M Spanish citizens and is the leading modifiable contributor to cardiovascular disease and death. Our society has already identified balanced diet, physical activity and emotional wellbeing as the 3 pillars of healthy living. Healthy sleep should be incorporated as the fourth pillar, as clearly supported by the extensively available scientific evidence. Targeting sleep is considered the new frontier in cardiovascular prevention. In fact, recent scientific evidence encourages consideration of including sleep disturbances in the top 10 potentially modifiable cardiovascular risk factors. Sleep-disordered breathing affect 30-80% of patients with hypertension. The personalized management of hypertension is challenging due to; i) the misclassification of hypertensive patients (affecting 1 out of 3 patients); ii) the lack of adequate treatment of high mortality risk hypertensive phenotypes today is an unmet clinical need; iii) unawareness of the impact of sleep-disordered breathing as a modifiable risk factor for hypertension. Importantly, the investigators already made the seminal observations showing that the treatment for sleep-disordered breathing reduces blood pressure in the hypertensive phenotypes with the highest mortality risk. Given the need for novel strategies to treat hypertension and, supported by our data, the investigators propose to study and treat sleep-disordered breathing to improve hypertension control. METASLEEP will go beyond current state-of the-art providing a new paradigm for the accurate hypertension classification and treatment. This project will open up a new avenue on the therapeutic potential of the management of sleep-disordered breathing in hypertension.

DETAILED DESCRIPTION:
This project aims to implement a new hypertension management system, which will include the monitoring and treatment of respiratory disorders during sleep. This new precision medicine-based management will be carried out in the Primary Care setting and will improve blood pressure control, the main risk factor for the leading cause of death worldwide: cardiovascular diseases.

The current model for managing patients with essential hypertension is based on deciding when to treat with measures that go beyond dietary and lifestyle interventions. Once it is decided to treat the patient pharmacologically, the ideal drug is decided and during follow-up whether it is necessary to change the treatment or not. This entire process is usually carried out by the Primary Care doctors. The hypertension specialist is usually reserved for difficult-to-control cases or patients with resistant hypertension. In the current model there is little communication between the different levels of care. In addition, the study of the SDB is carried out completely independently of this process. The METASLEEP project aims to change this work dynamic. The creation of the METASLEEP PC-node centralizes care for patients with hypertension in the Primary Care team (physician and nurse). The PC-node will evaluate the patient comprehensively, incorporating 24-hour ambulatory blood pressure monitoring as well as a sleep study. There will be coordination with the hypertension specialist for the management of complex cases and with the sleep unit specialist to support therapeutic decisions or management of patients with complex sleep apnea. Moreover, our project aims to incorporate the precision medicine techniques, such as the HIPARCO-score in the clinical management of hypertensive patients. Furthermore, the investigators aim to identify the best option that guarantees the best control in different clinical situations, with the greatest anticipation and with the fewest side effects, as well as with the greatest additional benefits and, finally, when to modify the treatment.

The METASLEEP project aims to contribute to the development of personalized medicine tools by identifying the molecular profile that enables to develop a non-invasive model with clinical utility. This model will contribute to the characterization of the patient that is vulnerable to the deleterious effects of OSA and who would benefit from OSA treatment to improve cardiovascular morbidity. The availability of an instrument based on a biomarker profile for risk stratification will help the physician to make therapeutic decisions in individuals with OSA and hypertension, contributing to the change of the current clinical management guidelines. Likewise, molecular tools can be developed to identify the profile of the patient that positively respond to CPAP treatment (in terms of blood pressure decrease). Finally, the investigators will obtain data that will evaluate the economic impact of the METASLEEP project. This cost-effectiveness analysis will be carried out from the perspectives of both, the SNS and the social perspective. Importantly, the investigators have planned a specific objective to define and calculate quantitatively, qualitative and cost-effectively the METASLEEP project, compared to the conventional current procedure.

The overall objective of the METASLEEP project is to establish a new paradigm in the treatment of hypertension through the management of sleep disordered breathing (SDB).

The specific objectives, are the following:

1. To implement the management of hypertension based on the presence of nocturnal hypertension and SDB (METASLEEP model).
2. To depict a singular cluster of circulating miRNAs (METASLEEP-score) in patients with nocturnal hypertension and SDB.
3. To characterize highly responder patients that would benefit from SDB treatment in terms of blood pressure control.
4. To implement in the clinical practice the use of the HIPARCO-score technology for the management of resistant hypertension.
5. To evaluate the feasibility and acceptability of the METASLEEP model for the comprehensive clinical management of hypertension based in the management of SDB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arterial hypertension who visit their primary care physician in one of the participating primary care centers.
* Signature of the informed consent.

Exclusion Criteria:

* Psycho-physical inability to complete questionnaires.
* Patients with very limiting chronic disease.
* Previous diagnosis of OSA or any other sleeping disorder
* Active treatment with CPAP.
* Fixed night shift worker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients atttending to their primary care center for the control of their arterial hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 1523 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in nocturnal blood pressure | At 6 and 18 months
  Change in nocturnal blood pressure at 6 and 18 months with respect to baseline (mean night-time)

SECONDARY OUTCOMES:
Identification of circulating miRNAs in patients with nocturnal hypertension and sleep disordered breathing. | 6 and 18 months
  Identification a specific singular cluster of circulating miRNAs in patients with nocturnal hypertension and sleep disordered breathing.
Epigenetic, proteomic and metabolomic/lipidomic phenotype characterization | 6 and 18 months
  Characterization of the epigenetic, proteomic and metabolomic/lipidomic phenotype of hypertensive highly responders to CPAP treatment
Clinic phenotype characterization | 6 months
  Characterization of the clinic phenotype of hypertensive highly responders to CPAP treatment
Changes induced by exosomes | 6 months
  Changes in morphological, functional and molecular promoted by exosomes isolated from selected patients.
Validation the HIPARCO-Score tool in an independent cohort, men with resistant hypertension, OSA and CPAP compliance (≥4h/night) | 2 years
  Analyse mRNA to validate de HIPARCO score
Creation of a predictive tool (like HIPARCO-Score) for women | 2 years
  Identify a plasma miRNA profile that predicts blood pressure response to CPAP treatment.
Cost-Effectiveness analyses between study groups and to compare the cost of health care utilization between two year before and after the starting of the study related to the study groups. | After 18 months of follow-up
  Only direct costs will be considered. Analysis will include an estimation of quality-adjusted life-years (QALYs) gained
Validation of the METASLEEP score | 2 years
  Identify specific miRNAs signature that would have the capability to identify patients with nocturnal hypertension, likely to exhibit a favorable blood pressure response to SDB treatment for the blood pressure control.
CPAP compliance at 6 and 18 months | 6 and 18 months
  Objective data to be downloaded from the CPAP device
Satisfaction at 6 and 18 months | 6 and 18 months
  Visual analog scale. The Satisfaction test is a self-reported outcome measure composed by 3 items which are measured by ten ranges. Scores range from 0 to 10, with higher scores indicating better satisfaction.
Changes in Epworth Sleepiness Scale (ESS) | 6 and 18 months
  Changes in Epworth Sleepiness Scale (ESS). The ESS test is a self-reported outcome measure composed by 8 items which examine diurnal somnolence. Scores range from 0 to 28, with higher scores indicating more sleepines.
Changes in Quality of life: Test EuroQol | 6 and 18 months
  Changes in Quality of life: Test EuroQol. The EuroQol test is a self-reported outcome measure composed by 5 items which examine five dimensions of health (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression) and each of them has three levels of severity (no problems, some problems or moderate problems, and severe problems). Scores range from 0 to 1, with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé Illa, MD, Principal Investigator — Spanish Respiratory Society (SEPAR)
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinilla L, Benitez ID, Moncusi-Moix A, Torres G, Casanovas-Salvatella O, Juez-Garcia I, Gracia-Lavedan E, Alonso-Fernandez A, Caballero-Eraso C, Cano-Pumarega I, Boira I, Egea C, Gonzalez M, Mediano O, Roncero A, Roche-Campo F, Sanchez-Quiroga MA, Chai-Coetzer CL, Sanchez-de-la-Torre M, Barbe F, de Batlle J; Spanish Sleep Network. Impact of Sleep-disordered Breathing Management in Primary Care on Systemic Hypertension Control: Protocol for the METASLEEP Implementation Trial. Open Respir Arch. 2025 Nov 17;8(1):100522. doi: 10.1016/j.opresp.2025.100522. eCollection 2026 Jan-Mar. PMID 41477672